CLINICAL TRIAL: NCT04806516
Title: Development of Adaptive Deep Brain Stimulation (aDBS) for the Treatment of Intractable Obsessive-Compulsive Disorder (OCD) Phase II Using Summit RC+S System With ECoG Paddles
Brief Title: Phase II Adaptive Deep Brain Stimulation for Obsessive-Compulsive Disorder
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: University of Pittsburgh (Other); Brown University (Other); Carnegie Mellon University (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Medtronic (Industry)
Responsible Party: Principal Investigator, Wayne Goodman MD, D. C. and Irene Ellwood Professor and Chair, Baylor College of Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 49155; 1UH3NS100549 (NIH); 49340 (Other Grant/Funding Number: BCM ID)
Record Dates: First submitted 2021-03-17; First posted 2021-03-19 (Actual); Last update posted 2025-08-18 (Actual); Status verified 2025-08

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: Deep Brain Stimulation (DBS); Treatment Resistant OCD; Intractable OCD; Obsessive Compulsive Disorder (OCD); Cognitive Behavior Therapy (CBT); Exposure and Response Prevention (ERP)
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Intervention Model Description: At the end of month 8 after DBS implant, all subjects will enter a one-month delayed onset withdrawal period in which the subject and Independent Evaluators are blinded to timing of discontinuation. See description below.
Who Masked: Participant, Outcomes Assessor
Masking Description: In all cases, the sequence will be as follows in one-week segments: 100% Active, 50% Active, Sham and Sham. Subjects will be seen weekly. Amplitude will be reduced by 50% at start of week 2 and turned off at start of week 3. Subjects will be told that DBS will be discontinued at some point during the 4 weeks. The purpose of the 50% initial reduction is to minimize rebound effects. The programmer (not the PI in this case) will be open to the design and perform "sham" activation. Relapse is defined as a 25% increase of the Y-BOCS over two consecutive visits compared to discontinuation baseline.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Summit RC+S DBS Implant for OCD (Experimental): All subjects will receive surgical implantation of RC+S DBS system with ECoG paddles
  Interventions: Device: Summit RC+S System with ECoG Paddles
- One Month Blinded Discontinuation Period (Experimental): The subject and Independent Evaluators are blinded to timing of discontinuation. In all cases, the sequence will be as follows in one-week segments: 100% Active, 50% Active, Sham and Sham. Subjects will be seen weekly. Amplitude will be reduced by 50% at start of week 2 and turned off at start of week 3. Subjects will be told that DBS will be discontinued at some point during the 4 weeks. The purpose of the 50% initial reduction is to minimize rebound effects. The programmer (not the PI in this case) will be open to the design and perform "sham" activation as described previously. Relapse is defined as a 25% increase of the Y-BOCS over two consecutive visits compared to discontinuation baseline
  Interventions: Other: One Month Blinded Discontinuation Period:

INTERVENTIONS:
Device: Summit RC+S System with ECoG Paddles — Summit RC+S System with ECoG Paddles consists of:
  * Olympus RC+S implantable pulse generator (IPG), Model B35300R: 2 per subject x 5 subjects = 10 units
  * Extension Leads, Model 37087: 2 per subject X 5 subjects = 10 units
  * DBS Leads, Model 3387: 2 per subject X 5 subjects = 10 units
  * Patient Therapy Manager (PTM), Model 4NR009: 1 per subject x 5 subjects = 5 units
  * Recharge Therapy Manager (RTM), Model 97755: 1 per subject x 5 subjects = 5 units
  * Clinician Telemetry Module (CTM), Model 4NR011: 1 per subject x 5 subjects = 5 units
  * Research Lab Programmer (RLP), Model 4NR010: 1 unit
  * Research Software Development Kit (RDK), Model 4NR013: 2 units
  * Subdural Quadripolar Paddle Lead, Model 09130: 2 per subject x 5 subjects = 10 units
  Other Names: Deep Brain Stimulation System; DBS; Summit RC+S
  Arms: Summit RC+S DBS Implant for OCD
Other: One Month Blinded Discontinuation Period: — The subject and Independent Evaluators are blinded to timing of discontinuation. In all cases, the sequence will be as follows in one-week segments: 100% Active, 50% Active, Sham and Sham. Subjects will be seen weekly. Amplitude will be reduced by 50% at start of week 2 and turned off at start of week 3. Subjects will be told that DBS will be discontinued at some point during the 4 weeks. The purpose of the 50% initial reduction is to minimize rebound effects. The programmer (not the PI in this case) will be open to the design and perform "sham" activation as described previously. Relapse is defined as a 25% increase of the Y-BOCS over two consecutive visits compared to discontinuation baseline.
  Arms: One Month Blinded Discontinuation Period

SUMMARY:
This research study is for participants that have been diagnosed with intractable Obsessive -compulsive disorder (OCD). OCD is a persistent and oftentimes disabling disorder marked by unwanted and distressing thoughts (obsessions) and irresistible repetitive behaviors. OCD affects 2-3% of the US population, and is responsible for substantial functional impairment and increased risk of early death.

The only established first-line treatments for OCD are cognitive-behavioral therapy (CBT) with exposure and response prevention and certain medications. About 30-40% of patients fail to respond and few experience complete symptom resolution. Up to 25% of patients have difficulty tolerating CBT and the risk of relapse after therapies remains large. For the most severe cases, neurosurgery (surgery in the brain), has long been the option of last resort.

In this study the investigators want develop an adaptive Deep Brain Stimulation (aDBS) system to use in subjects with intractable (hard to control) OCD. Deep brain stimulation (DBS) remains investigational for OCD patients and is not considered standard therapy. DBS involves the surgical implantation of leads and electrodes into specific areas of the brain, which are thought to influence the disease. A pack implanted in the chest, called the neurotransmitter, keeps the electrical current coursing to the brain through a wire that connects the neurotransmitter and electrodes. It is believed DBS may restore balance to dysfunctional brain circuitry implicated in OCD. The goal of this study is to enhance current approaches to DBS targeting in the brain and to use a novel approach to find a better and more reliable system for OCD treatment.

This current research protocol will focus on the completion of Phase II which will implant the RC+S system with ECoG paddles in 5 subjects.

DETAILED DESCRIPTION:
ENROLLMENT: A subject is considered enrolled upon signing informed consent and deemed eligible to be screened by the investigator. The informed consent process may include discussions with the patients family and referring clinician. Medical records that can be obtained will be carefully reviewed to determine adequacy of past treatments including Cognitive Behavioral Therapy (CBT).

A subject identification number will be assigned to each subject that signs consent. This number will be used to identify the subject and must be used on all study documentation related to that subject throughout the study.

SCREENING: Potential subjects meeting inclusion/exclusion criteria and willing to participate in the study as demonstrated by signing the informed consent will be enrolled in the study and undergo 2 screening visits (Visit 1 and Visit 2) spaced over an approximate 1 month period. Diagnostic and screening ratings are completed, followed by complete medical, neurological and neurosurgical evaluations. Final selection of candidates will be made by consensus of the multi-disciplinary investigator team (Project Advisory Committee).

Neuroimaging Methods:

The Core for Advanced MR Imaging (CAMRI) is a state-of-the-art resource housing 3 cutting edge MRI systems for the Houston research community, located at BCM Main Campus. CAMRI will perform the research 3T MRI scans, which will be collected on all subjects (DBS and control) using the Prisma scanner for consistency. All subjects will be escorted to CAMRI by the study team.

DBS implanted subjects will undergo two 3T MRI Scans prior to surgery (1 research MRI at CAMRI and 1 clinical MRI at Baylor St. Luke's Medical center (BSLMC). DBS implanted subjects will under 4 Magnetoencephalography (MEG) scans total.

Control subjects will undergo one 3T MRI scan (research MRI scan at CAMRI). Control subjects will also undergo 4 MEG scans.

TREATMENT: Subjects eligible for DBS implantation will also have an additional clinical, pre-surgical 3T MRI scan performed at baseline. This scan will be performed on a Philips scanner at Baylor St. Luke's Medical Center (BSLMC). This scan is necessary in order to potentially screen out individuals presenting with brain abnormalities which would not be compatible with the surgery (e.g., congenital defects, lack of normal anatomic correlates) and to assist with surgical planning.

All Subjects (DBS and control) will also undergo MEG scans. This is also needed as a baseline assessment as MEG scans will also be performed post implantation at 2 weeks, 6 months, and 12 months on a MEG scanner at the Texas Childrens Hospital in the Houston Medical Center.

Chest X-ray and EKG will also be performed on OCD subjects eligible for DBS.

Age/gender matched non-implanted subjects will serve as controls. They will undergo 1-research 3T MRI and 4 MEG scans using the same imaging protocol and at the same time points as OCD implant subjects to control for non-DBS effects on rs-fc.

1. Unless collected prior to the day of surgery, a head CT will be performed on the morning of surgery for stereotactic planning.
2. Employing local anesthetic (with or without sedation as clinically indicated), a stereotactic headframe (Leksell Model G, Elekta Instruments, Atlanta, GA, USA) will be attached to the subjects skull on the morning of surgery in the operating room.
3. A 3D volumetric image (O-Arm 2, Medtronic Inc, Boulder, CO, USA) will be performed for purposes of defining the volumetric stereotactic headspace.
4. The images will be uploaded onto a Computer Workstation (Stealth S7, Medtronic, Inc., Boulder, CO, USA) equipped with stereotactic planning software (Cranial 3.0) for the purpose of planning the surgery. The preoperative 3T MRI obtained prior to the surgical date, will be fused with the CT scan in the surgical planning station. The initial target point within the ventral striatum will be chosen based on the subjects specific anatomy. The surgical trajectory to this point will also be planned in order to avoid prominent vessels, the sulci, and the ventricles. The computer will generate the X, Y and Z coordinates to set on the frame as well as the coronal and sagittal angles of approach required to establish the desired trajectory and target point. This initial target point will be modified by the subjects specific anatomy as determined by the preoperative 3T scans. The final target coordinates will be determined during this analysis.
5. While the surgeon is planning the procedure, the subject will be positioned supine on the operating table. A Foley catheter will be inserted. Antibiotics will be administered intravenously and vital signs will be monitored. The stereotactic head frame will be fixed to the operating table for subject safety, with the head elevated for subject comfort. A sterile prep and drape will be performed.
6. The target coordinates will be set on the stereotactic frame bringing the target point to the center of the operating arc. Additional local anesthetic will be given at the point of incision. Following incision, a 14 mm burr hole will be made employing a self-stopping perforator. The burr hole cap provided with the DBS lead will be secured to the skull with two screws. The dura will be coagulated and incised. The pial surface will be gently coagulated and a small incision will be made to allow easy entry of the electrode guides, which will be inserted to the brain according to standard stereotactic protocol.
7. Once the above adjustments have been made, the DBS quadripolar electrode (model 3387; Medtronic Inc., Minneapolis, MN, USA) will be inserted through the guide tube to the target point. Reticles will be attached to the frame and intraoperative imaging will be employed to confirm that the lead tip is positioned at the target and assess for the presence of intracerebral hemorrhage. Sedation will be withdrawn. An extension cable will be connected to the lead sterilely and the other end will be passed off the field to be connected to an external pulse generator so that test stimulation may be performed. Test stimulation will be performed via each contact to 1) assess for stimulation-induced side effects and 2) monitor for acute changes in behavior using a Likert-type scale to assess anxiety, arousal, and mood. Intra operative behavioral testing of stimulation will be videotaped.
8. Phase II addition of ECoG. In order to achieve optimal coverage of the orbitofrontal cortex (OFC) region, the investigators will place a subdural cortical strip electrode over this region of cortex. There is well-established precedent for using strip electrodes over the OFC cortical surface, both in sub-acute (<1 month) and chronic (years/permanent) clinical settings. OFC strip electrodes have been commonly placed via a burr hole in the inferior frontal region for epilepsy monitoring. The electrodes used in these applications are usually 4 to 8 contacts, spaced 1 cm apart. These are typically sub-acute placements lasting days to weeks, and this practice has been common across the U.S. and world for decades. Strip electrodes covering OFC have also been used as permanent implants in the responsive neurostimulation (RNS) system, which is FDA approved and clinical standard of care for the treatment of medically refractory epilepsy. The strip electrodes used in this case are 4 contacts spaced 1 cm apart. In communications with the RNS device manufacturer, the investigators estimate that 100s of such electrodes have been placed in patients in this country. Our placement procedure will be very similar to that used for RNS OFC strip electrodes. The investigators will use the 09130 Subdural Quadripolar Paddle Lead, which is also 4 contacts spaced 1 cm apart. The investigators will create a burr hole in the inferior frontal region. The investigators will use standard frameless navigation to choose a location of the burr hole that facilitates a direct line of sight along the horizontal floor of the anterior cranial fossa within which lies the OFC region. The investigators will make a cosmetically acceptable incision approximately the same size as that used for the traditional DBS lead. The investigators will use monopolar cautery to deepen the incision past the temporalis muscle and create a standard size burr hole. The investigators will open the dura and visualize the inferior frontal lobe and floor of the anterior cranial fossa. Under direct vision, the investigators will place the strip electrode using irrigation to permit smooth placement, paying careful attention not to damage cortical vasculature. Bridging veins between dura and cortex are extremely rare in this region, thus increasing the safety profile of the procedure. Once the electrode is in place, the investigators will suture its tail to the dura in the burr hole to provide an anchor point. The investigators will then use a small metal plate to affix the electrode tail to the outer aspect of the skull near the burr hole to further anchor the electrode. The investigators will use a small length of plastic tubing available in the electrode kit as a shock absorber around the electrode tail at this fixation point to avoid chronic mechanical damage to the electrode tail from contact with the plate. The investigators place fibrin glue within the burr hole to prevent leak of cerebrospinal fluid. The investigators will close the muscle with dissolvable sutures, tunnel the tail to the DBS lead burr hole, and close the incision in standard fashion. From the site of the DBS lead burr hole, the two electrode tails (one for the DBS lead and the other for the OFC strip electrode) will be tunneled towards the ipsilateral IPG site in standard fashion.
9. Intra-operative X-ray imaging may be performed as needed (up to 4 times per side) to ensure proper target has been reached.
10. A post-implantation 3D volumetric scan will be performed to confirm the electrode position.
11. Steps 5-9 above will be performed to insert the second DBS lead and ECoG paddle in the other hemisphere to complete implantation of all electrodes.
12. If there are no untenable side effects, the leads will be secured to the skull with the burr hole caps. The free end of the leads will be left in the sub-galeal space and the incisions will be closed in anatomical layers.
13. The headframe will be removed and general anesthesia will be induced. Two Olympus RC+S pulse generators will then be implanted in the subclavicular region and connected to the deep brain and cortical leads via extension cables (two IPGs, each driving one cortical and one subcortical lead).
14. A post-operative CT scan will be performed prior to discharge to ensure that an intracerebral hemorrhage has not occurred.
15. The subject will be taken to the Recovery Room or the Neurosurgery ICU for post- operative monitoring (See below) and will be discharged from the hospital after at least one night of observation and when clinically stable. A Basic Metabolic Panel (BMP) may be run on the subject to confirm they are clinically stable.
16. The subject will return to the neurosurgery clinic (Visit 4) for post-operative evaluation according to normal clinical practice (approximately 1 week after surgery). The wounds will be inspected and the subjects neurological status will be assessed. Sutures will be removed.

DBS Programming:

Initially, a monopolar survey will be conducted with frequency set to 150 Hz and pulse width to 90 microseconds. Constant current amplitude will be used and increased in a step-wise fashion as tolerated and without exceeding current density upper limits. The constant current setting is particularly useful in the early weeks to months following surgery when impedances are still changing. In order to elicit a mirth response, amplitude needs to return to 0 microamps for about 30 seconds before testing the next increment. For example, if 2mA, C+1, 90usec, 150Hz is ineffective, then amplitude is reduced to 0mA for 30 seconds and then rapidly increased to 4mA, C+1-, 90usec, 150Hz. Soft start needs to be turned off. Bipolar settings will also be tested and need to be used during rsfMRI. DBS parameters will be optimized/adjusted based on clinical evaluation of mood and anxiety and to minimize side effects. The following observed effects will be recorded via a scale used in a past study: facial expression, nervousness, alertness, and positive or negative affect. Facial expression will be measured using the AFAR system. AFAR will measure the maximum intensity and velocity of the smile response in action units. Participants faces will be recorded on video as their stimulation is increased to elicit the mirth response. Changes in facial expression using facial muscles of orbicularis oris (muscle that encircles the mouth) zygomaticus (major and minor muscles of the angle of the mouth) will be recorded. This information will be used to train a classifier to recognize that stimulation intensity is too great. The investigators will also have the subject self-report on changes in mood, anxiety, energy and side effects.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent prior to any study specific procedures being performed
2. Male or female between ages 21 and 70;
3. At least a five-year history of treatment-refractory OCD that causes substantial subjective distress and impairment in functioning;
4. A primary diagnosis of OCD with Y-BOCS minimum score of 28;
5. Failed an adequate trial of at least three of the following SSRIs: Fluoxetine; fluvoxamine; citalopram; escitalopram; sertraline; paroxetine;
6. Failed or could not tolerate an adequate trial of clomipramine;
7. Failed augmentation of one or more of the aforementioned drugs with at least one of the following antipsychotics: haloperidol; risperidone; quetiapine; ziprasidone; aripiprazole;
8. Failed an adequate trial of CBT for OCD, defined as 25 hours of documented exposure and response prevention (ERP) by an expert therapist;
9. Stable psychotropic medical regimen for the month preceding surgery

Exclusion Criteria:

1. Inability or refusal to give informed consent.
2. Lifetime diagnosis of psychotic disorders such as schizophrenia;
3. Alcohol or substance abuse/dependence within 6 months, excluding nicotine;
4. Deemed at high risk of suicidal behavior or impulsivity, per clinical opinion assessments.
5. Any Neurological/Medical condition that makes the subject, in the opinion of the surgeon, a poor candidate.
6. Pregnant (confirmed by serum pregnancy test on females of child bearing age) or plans to become pregnant in the next 24 months.
7. Need for Diathermy
8. Contraindications to MRI
9. Contraindications to MEG
10. Subject is determined to not be appropriate for this study based on the medical expertise of the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Percent of subjects that display biomarkers of OCD-related distress | Month 6
  electrophysiological signals (deep brain local field potentials with electrocorticography) from the brain showing Cohen's kappa k > 0.40, chance corrected classification agreement with OCD-related distress during task exposure in clinic.
Percent of subjects that display biomarkers of OCD-related distress | Month 9
  electrophysiological signals (deep brain local field potentials with electrocorticography) from the brain showing Cohen's kappa k > 0.40, chance corrected classification agreement with OCD-related distress during task exposure in clinic.
Percent of subjects that display biomarkers of OCD-related distress | Month 12
  electrophysiological signals (deep brain local field potentials with electrocorticography) from the brain showing Cohen's kappa k > 0.40, chance corrected classification agreement with OCD-related distress during task exposure in clinic.
Percent of subjects that display biomarkers of OCD-related distress | Month 18
  electrophysiological signals (deep brain local field potentials with electrocorticography) from the brain showing Cohen's kappa k > 0.40, chance corrected classification agreement with OCD-related distress during task exposure in clinic.
Percent of subjects that display biomarkers of DBS-induced hypomania | Month 6
  electrophysiological signals (deep brain local field potentials with electrocorticography) from the brain showing Cohen's kappa k > 0.40, chance corrected classification agreement with DBS therapy during clinical visits.
Percent of subjects that display biomarkers of DBS-induced hypomania | Month 9
  electrophysiological signals (deep brain local field potentials with electrocorticography) from the brain showing Cohen's kappa k > 0.40, chance corrected classification agreement with DBS therapy during clinical visits.
Percent of subjects that display biomarkers of DBS-induced hypomania | Month 12
  electrophysiological signals (deep brain local field potentials with electrocorticography) from the brain showing Cohen's kappa k > 0.40, chance corrected classification agreement with DBS therapy during clinical visits.
Percent of subjects that display biomarkers of DBS-induced hypomania | Month 18
  electrophysiological signals (deep brain local field potentials with electrocorticography) from the brain showing Cohen's kappa k > 0.40, chance corrected classification agreement with DBS therapy during clinical visits.

SECONDARY OUTCOMES:
Change in Yale-Brown Obsessive Compulsive Scale (Y-BOCS) Rating OCD Symptom Severity | Baseline to 30 days
  Changes in the Yale-Brown Obsessive Compulsive Scale survey/questionnaire. This is measured after closed-loop stimulation and is an assessment to rate symptoms of OCD on a scale of 0-50 (with a higher number indicating a more severe outcome ratings of OCD and 0 indicated no symptoms of OCD).

CONTACTS AND LOCATIONS:
Overall Officials: Wayne Goodman, MD, Principal Investigator — Baylor College of Medicine
Locations (3):
- United States (3):
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Brown University, Providence, Rhode Island
  - Baylor College of Medicine, Houston, Texas